CLINICAL TRIAL: NCT01198379
Title: Efficacy of Monitoring of Aspirin Responsiveness in the Prevention of Cardiovascular Events and Decrease in Bleeding Complications in Patients With End-Stage Kidney Disease Undergoing Hemodialysis
Brief Title: Aspirin in the Prevention of Cardiovascular Events in Hemodialysis Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTCGHTN01
Record Dates: First submitted 2010-08-24; First posted 2010-09-10 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2018-01

CONDITIONS: End-Stage Renal Disease
Keywords: aspirin; aspirin resistance; hemodialysis; cardiovascular; Prevalence of aspirin resistance, cardiovascular events, and safety profile
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental)
  Interventions: Drug: aspirin
- Sugar pills (Placebo Comparator): Hemodialysis (HD) patients receive placebo not containing aspirin in this study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: aspirin — aspirin 100 mg qd for 3 years
  Arms: Aspirin
Drug: Placebo
  Arms: Sugar pills

SUMMARY:
The study is prospectively initiated to: (1) evaluate the alterations in platelet function to aspirin therapy and the prevalence of aspirin resistance in patients with chronic kidney disease undergoing hemodialysis, and (2) compare the incidence of vascular events (myocardial infarction, cardiac death, stroke, vascular access thrombosis, or revascularization procedure) and the safety profile among placebo-treated, aspirin-resistant and aspirin-sensitive patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with end-stage renal disease who are undergoing long-term hemodialysis.

Exclusion Criteria:

Patients will be excluded if there is evidence of

* a recent history of acute uremia,
* previous adverse reaction to a aspirin or history of aspirin hypersensitivity (eg, aspirin-induced asthma or angioedema),
* concurrent treatment with other antiplatelet agent (clopidogrel or ticlopidine), steroidal drugs, or nonsteroidal anti-inflammatory drugs,
* high immediate risk for bleeding (eg, active peptic ulceration, recent injury, or hemophilia), or
* life-threatening condition other than end-stage renal disease or vascular disease (eg, non-skin cancer).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02 (Estimated); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
the prevalence of aspirin resistance | 3 years

SECONDARY OUTCOMES:
the incidence of vascular events (myocardial infarction, cardiac death, stroke, vascular access thrombosis, or revascularization procedure) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Der-Cherng Tarng, MD, PhD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730